CLINICAL TRIAL: NCT01320527
Title: A Phase II Clinical Trial of a Vitamin/Nutriceutical Formulation for Alzheimer's Disease
Brief Title: A Clinical Trial of a Vitamin/Nutriceutical Formulation for Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Massachusetts, Lowell (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-1350; IIRG-08-91737
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: dietary supplement; cognition; mood; Alzheimer's disease; memory loss
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nutriceutical formulation (Experimental): Nutritional supplement
  Interventions: Dietary Supplement: Nutriceutical formulation
- Placebo 1 (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nutriceutical formulation — Two pills that collectively contain: folic acid (400µg), Vitamin B12 (6µg), Vitamin E (as alpha-tocopherol; 30 IU), S-adenosylmethionine (SAM; 400mg), N-acetyl cysteine (NAC; 600mg) and Acetyl-L-carnitine (ALCAR; 500mg). Taken once daily for duration of study (1 year).
  Other Names: MemoryXL
  Arms: Nutriceutical formulation
Other: Placebo — A mixture of 6 vitamins and nutriceuticals
  Arms: Placebo 1; Placebo 2

SUMMARY:
Based on prior published pilot studies, the investigators have initiated a larger, multi-site placebo-controlled clinical trial with Alzheimer's disease (AD) patients and individuals diagnosed with Mild Cognitive Impairment (MCI), with the hopes of (1) confirming (or denying) the above promising clinical findings, and (2) determining whether or not our formulation can delay MCI "conversion" to AD.

DETAILED DESCRIPTION:
Preclinical studies with mouse models of of age-related neurodegeneration led us to develop a Nutriceutical Formulation ("NF") consisting of 6 over-the-counter vitamins and nutriceuticals, that buffers multiple facets of Alzheimer's disease (AD), including (1) reducing presenilin expression, gamma-secretase activity, Abeta generation and tau phosphorylation, (2) buffering homocysteine and Abeta-induced oxidative damage, (3) reducing aggression, (4) increasing acetylcholine production and improving/maintaining cognitive performance.

A 1-year, open-label trial with NF with mild to moderate AD patients demonstrate improvement in cognitive performance (Dementia Rating Scale, Clock-drawing) within 3-6 months. Caregivers reported maintenance of daily performance and improved mood (ADCS-Activities of Daily Living and NeuroPsychiatric Inventory). A placebo-controlled study with moderate to late-stage AD indicates delayed cognitive decline and maintenance of daily activities. No adverse events were reported.

A multi-site trial with >90 individuals aged 45-73 without dementia indicated that NF statistically improved executive function (Trails B-A) vs. placebo within 3 months, which increased further at 6 months. The placebo group demonstrated identical improvement in a 3-month open-label extension. Following NF withdrawal, participants returned to baseline; statistically-significant improvement was restored once NF was individuals resumed.

We have initiated a larger, multi-site placebo-controlled clinical trial with AD patients and individuals diagnosed with Mild Cognitive Impairment (MCI), with the hopes of (1) confirming (or denying) the above promising clinical findings, and (2) determining whether or not our formulation can delay MCI "conversion" to AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or Mild Cognitive Impairment
* must be able to swallow pills

Exclusion Criteria:

* known or suspected bipolar disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
cognitive improvement or maintenance of cognitive performance | within 3 months of treatment
  Prior studies demonstrate cognitive improvement when treatment was initiated prior to or during mild-moderate Alzheimer's disease, and maintenance/ delayed decline in cognitive performance when treatment was initiated during moderate-severe Alzheimer's disease

SECONDARY OUTCOMES:
behavioral/psychotic symptoms | within 3 months after initiation of treatment
  Prior studies demonstrate improvement in mood and other behavioral symptoms when treatment was initiated during mild-moderate Alzheimer's disease, and maintenance/ delayed decline in mood and other behavioral symptoms when treatment was initiated during moderate-severe Alzheimer's disease

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Remington, Ph.D., Principal Investigator — UMass Lowell, Lowell, MA 01854
Locations (8):
- United States (8):
  - Naples Medical Center, Naples, Florida
  - University of Maryland, Baltimore, Maryland
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Rivercourt Residences, Groton, Massachusetts
  - Mary Immaculate Residential, Lawrence, Massachusetts
  - D'Youville Senior Care, Lowell, Massachusetts
  - Neurocognitive Institute, Mount Arlington, New Jersey
  - Advanced Memory Dynamics, Layton, Utah

REFERENCES:
- [Derived] Mota SI, Pita I, Aguas R, Tagorti S, Virmani A, Pereira FC, Rego AC. Mechanistic perspectives on differential mitochondrial-based neuroprotective effects of several carnitine forms in Alzheimer's disease in vitro model. Arch Toxicol. 2021 Aug;95(8):2769-2784. doi: 10.1007/s00204-021-03104-1. Epub 2021 Jun 24. PMID 34164711
- [Derived] Remington R, Bechtel C, Larsen D, Samar A, Page R, Morrell C, Shea TB. Maintenance of Cognitive Performance and Mood for Individuals with Alzheimer's Disease Following Consumption of a Nutraceutical Formulation: A One-Year, Open-Label Study. J Alzheimers Dis. 2016;51(4):991-5. doi: 10.3233/JAD-151098. PMID 26967219
- [Derived] Remington R, Bechtel C, Larsen D, Samar A, Doshanjh L, Fishman P, Luo Y, Smyers K, Page R, Morrell C, Shea TB. A Phase II Randomized Clinical Trial of a Nutritional Formulation for Cognition and Mood in Alzheimer's Disease. J Alzheimers Dis. 2015;45(2):395-405. doi: 10.3233/JAD-142499. PMID 25589719